CLINICAL TRIAL: NCT05856734
Title: Explore How Living Arrangements Impact Dietary Intake, Physical Activity, Sleep Patterns and Stress Levels, Which Contribute to Weight Gain in First-year Undergraduate Students at University of Aberdeen
Brief Title: Weight Gain in First-year University Students
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Ferdous Alharbi, Student, University of Aberdeen
Other Study IDs: SBSEC /09/2022/Sept
Record Dates: First submitted 2023-03-01; First posted 2023-05-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity
Keywords: freshman 15; weight gain; university students; first-year university students; stress; living arrangement; physical activity; dietary intake; alcohol consumption; weight change; sleep
MeSH Terms: conditions — Obesity; Weight Gain; Motor Activity; Alcohol Drinking; Body Weight Changes | interventions — Weights and Measures; Eating; Exercise Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- University students living at home: Group of university students
  Interventions: Device: Weight and body composition change; Behavioral: Change in dietary intake; Device: Change in physical activity; Behavioral: Change in stress; Behavioral: Change in socio-demographic characteristics; Device: Change in sleep
- University students living in private accommodation: Group of university students
  Interventions: Device: Weight and body composition change; Behavioral: Change in dietary intake; Device: Change in physical activity; Behavioral: Change in stress; Behavioral: Change in socio-demographic characteristics; Device: Change in sleep
- University students living in the halls of residence: Group of university students
  Interventions: Device: Weight and body composition change; Behavioral: Change in dietary intake; Device: Change in physical activity; Behavioral: Change in stress; Behavioral: Change in socio-demographic characteristics; Device: Change in sleep
- Non-university participants living in Aberdeen: Group of age-matched volunteers living in the same city
  Interventions: Device: Weight and body composition change; Behavioral: Change in dietary intake; Device: Change in physical activity; Behavioral: Change in stress; Behavioral: Change in socio-demographic characteristics; Device: Change in sleep

INTERVENTIONS:
Device: Weight and body composition change — 1- Anthropometric Measurements: Body Weight (BW), Body Mass Index (BMI), Sitting Height Ratio (SHR), Waist to Hip Ratio (WHR), Finger Ratio (FR), Body Fat (BF%), and Weight-for-age growth charts. (Single measure)
Behavioral: Change in dietary intake — 1. 24-hour recalls using Intake24 (online survey) over 3-day.
  2. Self reported questionnaire. (Single measure)
Device: Change in physical activity — 1. ActiGraph GT9X Link accelerometer over 7-day.
  2. Self reported questionnaire. (Single measure)
  Other Names: Behavioral
Behavioral: Change in stress — 1- Self reported questionnaire. (Single measure)
Behavioral: Change in socio-demographic characteristics — 1- Self reported questionnaire. (Single measure)
Device: Change in sleep — ActiGraph GT9X Link accelerometer over 7-day. (Single measure)

SUMMARY:
The transition to university from secondary school comes with many changes to living arrangements, dietary and alcohol intake, physical activity, and stress. The purpose of this study is to explore weight gain in new university students in the UK under the 'Freshman15' phenomenon. This phenomenon is an expression commonly used in the United States and Canada to describe a weight gain of 15 lbs (6.8 kg) in students who transition from secondary school to university life. The research will assess to investigate the impact of lifestyle factors that predict students' weight gain during their first year at the University of Aberdeen. The study specifically focuses on how these factors vary based on their living arrangement. Also, the change in lifestyle will be explored in relation to age-matched individuals not-attending The transition to university from secondary school comes with many changes to living arrangements, dietary and alcohol intake, physical activity, and stress. The purpose of this study is to explore weight gain in new university students in the UK under the 'Freshman15' phenomenon. This phenomenon is an expression commonly used in the United States and Canada to describe a weight gain of 15 lbs (6.8 kg) in students who transition from secondary school to university life. First aim: To investigate the impact of lifestyle factors that predict students' weight gain during their first year at the University of Aberdeen. The study specifically focuses on how these factors vary based on their living arrangement. Also, the change in lifestyle will be explored in relation to age-matched individuals not-attending university. Second aim: To examine changes in weight, living arrangements, dietary intake, physical activity, sleep and stress after one year at university with previous participation students who moved to their second year to understand the influence that university life has on these trends compared to their first visit at the beginning of their first year at the university.

DETAILED DESCRIPTION:
Detailed Description:

Recruitment will take place over two academic years using flyers sent via email or distributed face-to-face among undergraduate first-year students at the University of Aberdeen (e.g., the Freshers Week), as well as in different public areas, such as supermarkets and shopping centres. If participants agree to participate in this study by signing the consent form, their involvement will last around eight months.

Aim1 "Transition to university study" During each academic year, I will conduct three visits with participants: At the beginning of the academic year in late September/October (Visit 1), after 3 months in January (Visit 2), and after 8 months at the end of the academic year in mid-April/May (Visit 3).

The study will be an observational study with four groups including three groups of university student and a group of age-matched volunteers living in the same city that are not attending university as a control:

1. University students living at home.
2. University students living in private accommodation.
3. University students living in the halls of residence.
4. Non-university participants living in Aberdeen.

Aim 2 "Follow-up study" I will conduct one visit with previous participating students in the study 1: in September/October year, after one year at the university (Visit 4).

Participants will be asked to come to a designated room at the University of Aberdeen. Each appointment will be in the morning (approx. 15 to 30 minutes for each visit).

During each visit, participants will be provided with further details concerning the study and given time to ask questions.

Measures:

1. Anthropometric Measurements will be taken: Body Weight (BW), Body Mass Index (BMI), Sitting Height Ratio (SHR), Waist to Hip Ratio (WHR), Finger Ratio, Body Fat (BF%), and Weight-for- Age Growth Charts.
2. Dietary intake will be examined in two distinct ways. Firstly, self reported questionnaire. Secondly, participants will be asked to complete 3 * 24-hour recalls to assess their consumption of ( protein (g), fat (g), carbohydrate (g), energy (kJ), alcohol (g), total sugars (g), non milk extrinsic sugars (g), fruit (g), vegetable (g), meat (g), processed meat (g), poultry (g), and fish (g) ). They will report two weekdays and one weekend day by using Intake24 online dietary recall system.
3. Physical activity will be examined in two ways. Firstly, self reported questionnaire. Secondly, participants will use an ActiGraph GT9X Link accelerometer (placed on the waist) to assess their physical activity (h), Activity intensity level (min).
4. Sleep patterns will be examined by ActiGraph GT9X Link accelerometer (placed on the waist) to assess their total awake duration (min), total sleep duration(min), bedtime (hh:mm), and wake time (hh:mm).
5. Stress: will be assessed via self reported questionnaire.
6. Socio-demographic characteristics: will be assessed via self reported questionnaire.
7. Changes in lifestyle behaviours: will be assessed via self reported questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Full-time first-year undergraduate students attending the University of Aberdeen or age-matched non-university participants living in Aberdeen.
* Aged between 17-20 years old.
* Both males and females will be recruited.

Exclusion Criteria:

* Over 20 years old,
* Pregnant/lactating, or taking medication which may affect their weight.

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: About 80 participants will be either full-time first-year undergraduate students attending the University of Aberdeen or age-matched non-university participants living in Aberdeen. Participants will be aged between 17-20 years. Both males and females will be recruited. Participants for the University categories will be recruited from across the range of programmes and living in (1) halls of residence (2) private accommodation (3) remaining at the family home. They may be UK or international students. The non-university volunteers may live in the family home or out of the home but must be recent high school graduates (within two years of graduating)
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight (BW) | Baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Weight (kilograms) will be measured using a Bioimpedance (Tanita MC-580 P).
Change in Body Mass Index (BMI) | Baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Body Mass Index (BMI) will be measured height (Metres) using a Stadiometer and body weight (kilograms) using a Bioimpedance (Tanita MC-580 P). BMI (kg/m2) will be calculated by dividing weight by height squared.
Change in Waist to Hip Ratio (WHR) | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Waist to Hip Ratio (WHR) is the ratio of waist circumference to the hip circumference will be measured using tape (CM) . WHR will be calculated as WC divided by HC.
Change in Body Fat (BF%) | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Body Fat (BF%) will be measured by Bioimpedance (Tanita MC-580 P).
Change in Weight-for- Age Growth Charts | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Weight-for- Age Growth Charts will be used to calculate the weight for age percentile, and this done by calculator using this website (the Center for Disease Center (CDC) children charts for 2-20 year olds). Weight for age percentile will be calculated by entering (gender, birthday, weight, and measurement date).
Change in Finger Ratio | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Finger Ratio will be measured using Vernier Caliper. I will measure the length of participant's index finger 2D of right hand from crease to tip. Then do the same for the ring finger 4D. Finger Ratio will be calculated as index finger 2D /ring finger 4D.

SECONDARY OUTCOMES:
Change in Protein Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Protein intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for protein intake (g)
Change in Fat Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Fat intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for fat intake (g)
Change in Carbohydrate Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Carbohydrate intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for carbohydrates intake (g)
Change in Energy Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Energy intake (kJ) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for energy intake (kJ)
Change in Alcohol Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Alcohol intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for alcohol intake (g)
Change in Total Sugars Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Total sugars intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for total sugars intake (g)
Change in Non-milk Extrinsic Sugars Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Non-milk extrinsic sugars intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for non-milk extrinsic sugars intake (g)
Change in Fruit Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Fruit intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for fruit intake (g)
Change in Vegetable Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Vegetable intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for vegetable (g)
Change in Meat Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. meat intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for meat intake (g)
Change in Processed Meat Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Processed meat intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for processed meat intake (g)
Change in Poultry Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Poultry intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for poultry intake (g) to assess change from baseline to follow-up after three months and at eight months.
Change in Fish Intake using intake24 | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete 3 * 24-hour recalls recording. Fish intake (g) will be calculated as follows: day 1= sum, day 2= sum, and day 3=sum, after that I will calculate the average of the three days for fish intake (g)
Change in Dietary Intake using questionnaire | Baseline at the beginning of the academic year, then a follow-up after three months, and at eight months (end of the academic year ).
  Participants will be asked to complete a questionnaire. It includes six multiple-choice questions to evaluate dietary behaviours. I have categorical data with repeated measures, so I will use non parametric analysis with repeated measures to assess change from baseline to follow-up after three months and at eight months.
  The first question require participants to report their daily calorie intake to maintain their current weight or to lose weight (such as yes, I have been for six months or longer/yes, I have but for less than six months/no, but I intend to in the next 30 days/no, but I intend to in the next six months/no, and I do not intend to in the next six months) etc.
Change in Physical Activity on Weekdays using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will wear ActiGraph GT9X Link accelerometers for seven consecutive days. To calculate hourly physical activity, the vector magnitude (VM) data for each minute within an hour (specifically, from 0:00 to 0:59 etc.) will summed. Subsequently, the average hourly physical activity (PA) will computed by considering the days when the monitor was worn.
Change in Physical Activity on Weekends using ActiGraph. | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will wear ActiGraph GT9X Link accelerometers for seven consecutive days. To calculate hourly physical activity, the vector magnitude (VM) data for each minute within an hour (specifically, from 0:00 to 0:59 etc.) will summed. Subsequently, the average hourly physical activity (PA) will computed by considering the days when the monitor was worn.
Change in activity intensities using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  To calculate the average activity counts per minute and the percentages of time spent in different activity intensities (sedentary, light, moderate, vigorous, and very vigorous), Actilife software version 6.13.4 will used. The analysis incorporate the use of the Freedson Adult 1998 cut-off points with an epoch length of 60 seconds.
Change in Total Awake Duration on weekdays using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will wear ActiGraph GT9X Link accelerometers for seven consecutive days. I will collected total awake duration (min) on weekdays (day 1= sum, day 2= sum, day 3=sum, and day 4= sum after that the average of four days will be collected)
Change in Total Awake Duration on Weekends using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will wear ActiGraph GT9X Link accelerometers for seven consecutive days. I will collected total awake duration (min) on weekends (day 1 = sum and day 2 = sum after that the average of two days will be collected)
Change in Total Sleep Duration on Weekdays using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will wear ActiGraph GT9X Link accelerometers for seven consecutive days. I will collected total sleep duration (min) on weekdays (day 1= sum, day 2= sum, day 3=sum, and day 4= sum after that the average of four days will be collected)
Change in Total Sleep Duration on Weekends using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will wear ActiGraph GT9X Link accelerometers for seven consecutive days. I will collected total sleep duration (min) on weekends (day 1 = sum and day 2 = sum after that the average of two days will be collected)
Change in Bedtime on Weekdays using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Bedtime will determine by identifying sudden periods of decreased activity levels which will dropped to zero and remained at that level for at least 5 consecutive epochs. To gain a metric variable, hours will count from 0 to 24, and hours after midnight will be counted as 25 (for 1:00), 26 (for 2:00), and so forth, which will then converted to decimal form; for instance, a bedtime of 21:30 will code as 9.50. The average bedtime will be analysed in hours and minutes (hh:mm) format.
Change in Bedtime on Weekends using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Bedtime will determine by identifying sudden periods of decreased activity levels which will dropped to zero and remained at that level for at least 5 consecutive epochs. To gain a metric variable, hours will count from 0 to 24, and hours after midnight will be counted as 25 (for 1:00), 26 (for 2:00), and so forth, which will then converted to decimal form; for instance, a bedtime of 21:30 will code as 9.50. The average bedtime will be analysed in hours and minutes (hh:mm) format.
Change in Wake Time on Weekdays using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Wake time will identify by finding the first epoch of sustained high activity (over 10 activity counts) after a period of at least five 30-second epochs with less than 10 activity counts. To gain a metric variable, hours will count from 0 to 24, and hours after midnight will count as 25 (for 1:00), 26 (for 2:00), and so forth, which will then converted to decimal form; for instance, a wake time of 07:39 will code as 7.65. The average wake time will be analysed in hours and minutes (hh:mm) format.
Change in Wake Time on Weekends using ActiGraph | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Wake time will identify by finding the first epoch of sustained high activity (over 10 activity counts) after a period of at least five 30-second epochs with less than 10 activity counts. To gain a metric variable, hours will count from 0 to 24, and hours after midnight will count as 25 (for 1:00), 26 (for 2:00), and so forth, which will then converted to decimal form; for instance, a wake time of 07:39 will code as 7.65. The average wake time will be analysed in hours and minutes (hh:mm) format.
Change in Physical Activity using questionnaire. | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Participants will be asked to complete a questionnaire that will evaluate physical activity. It includes six multiple-choice questions. I have categorical data with repeated measures, so I will use non parametric analysis with repeated measures to assess change from baseline to follow-up after three months and at eight months.
  For example, physical activity will assessed by asked participants to report which best describes their level of physical activity (e.g., I am inactive and don't plan on starting in the next six months/ I am inactive but I'm thinking about starting in the next six months/ I do a bit of physical activity, but not a lot/ I have been doing physical activity for six months/ I have been doing physical activity for more than six months) etc.
Change in Stress using questionnaire | baseline at the beginning of the academic year, then a follow-up after three months, at eight months (end of the academic year ), and after one year.
  Stress will be assessed by employing a questionnaire which evaluates stress levels in the students. It includes four multiple-choice questions. I have categorical data with repeated measures, so I will use non parametric analysis with repeated measures to assess change from baseline to follow-up after three months and at eight months.
  For example, the first question will asked participants to answer with (Yes /No) "Are you comfortable at their present level of stress?". The second question will, "How often do you feel stress?" participants provided with these options to choose from (e.g., (always/sometimes/rarely/never) etc..
Change in lifestyle behaviours using questionnaire | After one year at university
  lifestyle behaviours will be assessed by employing a questionnaire which evaluates changes in lifestyle behaviours. It includes eleven multiple-choice questions. I have categorical data with repeated measures, so I will use non parametric analysis with repeated measures to assess change after one year at university.
  for example, the first question will asked participants to answer with (Yes /No) "Do you still live in the same place?".
  Question 2. "Living Arrangement" (Home with family/Private accommodation/Halls of residence)3 Question 3. " Do you believe your eating habits have changed since the start of university?" (Yes/ No) etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes